CLINICAL TRIAL: NCT04794322
Title: Ovarian Cancer Detection by Uterine Lavage DNA and Serum Proteins: a Phase 2 Biomarker Study
Brief Title: Developing a Test of Uterine Lavage for the Detection of Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other); Fred Hutchinson Cancer Center (Other); Anne Arundel Health System Research Institute (Other); University of Arkansas (Other); National Cancer Institute (NCI) (NIH); Kaiser Permanente (Other); McGill University (Other); M.D. Anderson Cancer Center (Other); Swedish Medical Center (Other); Early Detection Research Network (Network)
Responsible Party: Principal Investigator, Steven Skates, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 20-450; 5U01CA152990 (NIH); U2CCA271871 (NIH)
Record Dates: First submitted 2021-02-19; First posted 2021-03-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Neoplasms; Ovarian Epithelial Carcinoma; Fallopian Tube Neoplasms; High Grade Ovarian Serous Adenocarcinoma; Stage I Ovarian Cancer; Stage II Ovarian Cancer; Stage III Ovarian Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8
Keywords: Uterine Lavage; Tumor DNA; Serum proteins; Ovarian neoplasms; Ovarian epithelial carcinoma; Ovarian cancer; Ovarian epithelial cancer; Neoplasms; Ovarian diseases; Early detection
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Neoplasms; Ovarian Diseases | interventions — Blood Specimen Collection; Papanicolaou Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Serum (red-top tubes)
  * EDTA plasma (purple-top tubes)
  * Uterine Lavage supernatant (conical tube)
  * Uterine Lavage filter (conical tube)
  * Uterine Lavage cell pellet (conical tube)
  * Buffy coat (purple-top tubes)
  * Tissue sections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pelvic Mass Cohort (cohort #1): 200 participants scheduled for surgery for suspected ovarian cancer due to a pelvic mass but without a confirmed tissue or cytology diagnosis.
  Interventions: Diagnostic Test: Uterine lavage, or a wash of the womb; Diagnostic Test: Blood sample; Diagnostic Test: Pap smear
- BRCA1/2 Carriers Cohort (cohort #2): 50 participants with an inherited BRCA1 or BRCA2 deleterious mutation without suspected ovarian cancers who are scheduled for risk-reducing salpingo-oophorectomy (RRSO) to remove ovaries and fallopian tubes.
  Interventions: Diagnostic Test: Uterine lavage, or a wash of the womb; Diagnostic Test: Blood sample; Diagnostic Test: Pap smear

INTERVENTIONS:
Diagnostic Test: Uterine lavage, or a wash of the womb — Uterine lavage is performed during surgery using a flexible, 3-way balloon tipped catheter. The catheter is inserted through the cervix, the balloon expanded and the uterine cavity lavaged using 10 cc of sterile saline which is collected, processed and stored for later analysis.
Diagnostic Test: Blood sample — Participants undergo two blood draws (one required, one optional) up to 31 days before surgery
Diagnostic Test: Pap smear — Participants undergo a standard Papanicolaou smear to collect cells and fluid from the cervix.

SUMMARY:
The study aims to develop a test for early detection of ovarian cancer using DNA from a growth involving the ovary found in a washing of the uterus (womb), and proteins found in the blood. The samples of the wash and the blood will be taken before surgery. After surgery, doctors will determine whether the participant had ovarian cancer or a benign disease of the ovaries. The tests of the washings and the blood will be examined to see how much the participants with ovarian cancer can be separated from the participants with a benign ovarian disease by the tests. Small amounts from the washing and the blood samples will be sent to four sites for analysis.

Statistical analyses of these data will compare tumor DNA found in the washing of the uterus with proteins in the blood to detect cases of ovarian cancer. The primary goal is to find tests that are mostly positive for cases of ovarian cancer and mostly negative for patients with benign disease. It is hoped that if the tests work for participants with symptoms of the disease that these tests will also work when testing women who have no symptoms. A new study would be needed to see if the tests worked in this situation. If the tests work, this could lead to increasing the number of cases detected in early stage disease and decreasing the number of cases detected in late stage disease. If this change in late stage is large, it will likely reduce deaths due to ovarian cancer.

DETAILED DESCRIPTION:
The study aims to elucidate the relative contributions to detection of ovarian cancer from tumor DNA in uterine lavage (UL) and protein biomarkers from blood using newly available detection and sample collection technologies. In this document, the term "ovarian cancer" includes fallopian tube cancer. In the first cohort, the study will enroll 200 participants. Enrolling participants prior to surgical diagnosis (e.g. laparoscopy or paracentesis) ensures the study will be "Prospective Collection of Samples, Blinded Evaluation" (PRoBE) compliant. The expectation is that ~50 of these participants will have pathologically confirmed ovarian cancer. In a second cohort, 50 participants will be enrolled. Based on published reports, it is expected that ~5 participants will have microscopic or low volume ovarian cancer. In each cohort, the participants with a pathologic invasive epithelial ovarian cancer diagnosis will be defined as Cases and participants without any ovarian cancer, primary peritoneal cancer (PPC), or other cancer identified due to the surgery, will be defined as Controls. Other cancer groups are: (i) PPC, (ii) non-invasive serous tubal intraepithelial carcinoma (STIC) lesions, (iii) non-epithelial ovarian cancers, and (iv) non-ovarian cancers.

Two sites will sequence DNA obtained from uterine lavages to detect tumor-derived DNA (tDNA): one will carry out Duplex Sequencing of TP53 and the second site will carry out Haloplex sequencing of an 18-gene panel. Two other sites will assay serum proteins: the first will use clinical grade assays for CA125 and HE4, and the second will use research grade assays for these two proteins plus four additional protein biomarker candidates. Statistical analyses of these data will evaluate the relative utility of tDNA and plasma proteins to detect Cases (sensitivity) while limiting detection of Controls (specificity) in these two cohorts. Remaining DNA from UL and blood based biospecimens in form of plasma, serum, and buffy coat will be stored at a biorepository at NCI Frederick for future biomarker investigations which include (but are not limited to) other methods of detecting tDNA from UL, tDNA from plasma, exosomal markers, and additional blood-based and UL biomarker candidates.

Primary objectives:

1. To collect samples from 200 participants with suspected ovarian cancer (of which ~50 or more are expected to have pathologically confirmed ovarian cancer) and 50 participants undergoing a risk-reducing salpingo-oophorectomy (of which ~5 are expected to have microscopic or low volume ovarian cancer).
2. To test the tDNA from uterine lavage samples for tumor-derived TP53 mutations, using Duplex sequencing, and for potential abnormalities in an 18-gene panel, using Haloplex sequencing
3. To test the serum proteins with two assays: the first will use clinical grade assays for CA125 and HE4, and the second will use research grade assays for these two proteins plus four additional protein biomarker candidates.

Outline: Participants undergo two blood draws (one required, one optional) up to 31 days before surgery and a uterine lavage at the time of planned surgery. The tDNA and serum proteins are then extracted from the samples and sent for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Has intact uterus (no history of uterine ablation, tubal ligation or bilateral salpingectomy)
* Cohort 1 (n=200 participants): Women scheduled for surgery or diagnostic laparoscopy for suspected but undiagnosed ovarian/fallopian tube cancer
* Cohort 2 (n=50 participants): Known BRCA1 or BRCA2 mutation carrier scheduled for risk-reducing salpingo-oophorectomy

Exclusion Criteria:

* Current tissue or cytology diagnostic procedure positive for ovary cancer or any cancer
* Inability to provide informed consent
* Age less than 30 years
* Inability to obtain the minimum amount of blood
* Inability to obtain the minimum amount of uterine lavage sample
* At risk if blood were drawn (e.g. hemophilia, serious anemia- Hb less than 8.0 gm/dL)
* Prior history of known ovarian or endometrial cancer
* Treatment less than 1 year (excluding hormonal therapy) for cancer that spread beyond its origin
* History of untreated high-grade cervical dysplasia (CIN3)
* History of treated high grade cervical dysplasia (CIN3) with a cytologically abnormal pap smear within the past year. If there is no post treatment Pap smear in the medical record, perform a Pap smear prior to the day of surgery. If this Pap smear is abnormal, the participant is ineligible.
* Currently pregnant
* Known Lynch syndrome

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohorts will be selected from patients scheduled for ovarian disorder-related surgeries across six sites: Massachusetts General Hospital in Boston, Massachusetts; Luminis Health System in Annapolis, Maryland; Johns Hopkins University School of Medicine in Baltimore, Maryland; Kaiser Permanente - San Francisco in San Francisco, California; the Swedish Medical Center in Seattle, Washington; and the University of Arkansas for Medical Sciences in Little Rock, Arkansas.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Genomic biomarkers assessing mutations and methylation of tumor DNA, and protein biomarkers measured as the concentration of a protein in pg/mL, both types of biomarkers measured in the collected biospecimens. | From enrollment through to pathology results post-surgery (usually same day)
  Biomarkers that distinguish between ovarian cancer and benign ovarian disease

CONTACTS AND LOCATIONS:
Overall Officials: Christos Patriotis, PhD, Study Director — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente - San Francisco, San Francisco, California
  - Anne Arundel Health System, Annapolis, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Swedish Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not anticipated to be shared.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Jacobs IJ, Menon U, Ryan A, Gentry-Maharaj A, Burnell M, Kalsi JK, Amso NN, Apostolidou S, Benjamin E, Cruickshank D, Crump DN, Davies SK, Dawnay A, Dobbs S, Fletcher G, Ford J, Godfrey K, Gunu R, Habib M, Hallett R, Herod J, Jenkins H, Karpinskyj C, Leeson S, Lewis SJ, Liston WR, Lopes A, Mould T, Murdoch J, Oram D, Rabideau DJ, Reynolds K, Scott I, Seif MW, Sharma A, Singh N, Taylor J, Warburton F, Widschwendter M, Williamson K, Woolas R, Fallowfield L, McGuire AJ, Campbell S, Parmar M, Skates SJ. Ovarian cancer screening and mortality in the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS): a randomised controlled trial. Lancet. 2016 Mar 5;387(10022):945-956. doi: 10.1016/S0140-6736(15)01224-6. Epub 2015 Dec 17. PMID 26707054
- [Background] Skates SJ. Ovarian cancer screening: development of the risk of ovarian cancer algorithm (ROCA) and ROCA screening trials. Int J Gynecol Cancer. 2012 May;22 Suppl 1(Suppl 1):S24-6. doi: 10.1097/IGC.0b013e318256488a. PMID 22543916
- [Background] Skates SJ, Greene MH, Buys SS, Mai PL, Brown P, Piedmonte M, Rodriguez G, Schorge JO, Sherman M, Daly MB, Rutherford T, Brewster WR, O'Malley DM, Partridge E, Boggess J, Drescher CW, Isaacs C, Berchuck A, Domchek S, Davidson SA, Edwards R, Elg SA, Wakeley K, Phillips KA, Armstrong D, Horowitz I, Fabian CJ, Walker J, Sluss PM, Welch W, Minasian L, Horick NK, Kasten CH, Nayfield S, Alberts D, Finkelstein DM, Lu KH. Early Detection of Ovarian Cancer using the Risk of Ovarian Cancer Algorithm with Frequent CA125 Testing in Women at Increased Familial Risk - Combined Results from Two Screening Trials. Clin Cancer Res. 2017 Jul 15;23(14):3628-3637. doi: 10.1158/1078-0432.CCR-15-2750. Epub 2017 Jan 31. PMID 28143870
- [Background] Rosenthal AN, Fraser LSM, Philpott S, Manchanda R, Burnell M, Badman P, Hadwin R, Rizzuto I, Benjamin E, Singh N, Evans DG, Eccles DM, Ryan A, Liston R, Dawnay A, Ford J, Gunu R, Mackay J, Skates SJ, Menon U, Jacobs IJ; United Kingdom Familial Ovarian Cancer Screening Study collaborators. Evidence of Stage Shift in Women Diagnosed With Ovarian Cancer During Phase II of the United Kingdom Familial Ovarian Cancer Screening Study. J Clin Oncol. 2017 May 1;35(13):1411-1420. doi: 10.1200/JCO.2016.69.9330. Epub 2017 Feb 27. PMID 28240969
- [Background] Maritschnegg E, Wang Y, Pecha N, Horvat R, Van Nieuwenhuysen E, Vergote I, Heitz F, Sehouli J, Kinde I, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Speiser P, Zeillinger R. Lavage of the Uterine Cavity for Molecular Detection of Mullerian Duct Carcinomas: A Proof-of-Concept Study. J Clin Oncol. 2015 Dec 20;33(36):4293-300. doi: 10.1200/JCO.2015.61.3083. Epub 2015 Nov 9. PMID 26552420
- [Background] Krimmel JD, Schmitt MW, Harrell MI, Agnew KJ, Kennedy SR, Emond MJ, Loeb LA, Swisher EM, Risques RA. Ultra-deep sequencing detects ovarian cancer cells in peritoneal fluid and reveals somatic TP53 mutations in noncancerous tissues. Proc Natl Acad Sci U S A. 2016 May 24;113(21):6005-10. doi: 10.1073/pnas.1601311113. Epub 2016 May 5. PMID 27152024
- [Background] Risques RA, Kennedy SR. Aging and the rise of somatic cancer-associated mutations in normal tissues. PLoS Genet. 2018 Jan 4;14(1):e1007108. doi: 10.1371/journal.pgen.1007108. eCollection 2018 Jan. PMID 29300727
- [Background] Gilbert L, Basso O, Sampalis J, Karp I, Martins C, Feng J, Piedimonte S, Quintal L, Ramanakumar AV, Takefman J, Grigorie MS, Artho G, Krishnamurthy S; DOvE Study Group. Assessment of symptomatic women for early diagnosis of ovarian cancer: results from the prospective DOvE pilot project. Lancet Oncol. 2012 Mar;13(3):285-91. doi: 10.1016/S1470-2045(11)70333-3. Epub 2012 Jan 17. PMID 22257524
- [Background] Cancer Genome Atlas Research Network. Integrated genomic analyses of ovarian carcinoma. Nature. 2011 Jun 29;474(7353):609-15. doi: 10.1038/nature10166. PMID 21720365
- [Background] Kinde I, Bettegowda C, Wang Y, Wu J, Agrawal N, Shih IeM, Kurman R, Dao F, Levine DA, Giuntoli R, Roden R, Eshleman JR, Carvalho JP, Marie SK, Papadopoulos N, Kinzler KW, Vogelstein B, Diaz LA Jr. Evaluation of DNA from the Papanicolaou test to detect ovarian and endometrial cancers. Sci Transl Med. 2013 Jan 9;5(167):167ra4. doi: 10.1126/scitranslmed.3004952. PMID 23303603
- [Background] Pepe MS "The Statistical Evaluation of Medical Tests for Classification and Prediction". Oxford University Press (2003)
- [Background] Gilbert L, Revil T, Meunier C, Jardon K, Zeng X, Martins C, Arseneau J, Fu L, North K, Schiavi A, Ehrensperger E, Artho G, Lee T, Morris D, Ragoussis J. The empress of subterfuge: cancer of the fallopian tube presenting with malapropism. Lancet. 2017 Sep 2;390(10098):1003-1004. doi: 10.1016/S0140-6736(17)31586-6. No abstract available. PMID 28872014
- [Derived] Greenwood A, Woodruff ER, Nguyen C, Piper C, Clauset A, Brubaker LW, Behbakht K, Bitler BG. Early Ovarian Cancer Detection in the Age of Fallopian Tube Precursors: A Systematic Review. Obstet Gynecol. 2024 Mar 1;143(3):e63-e77. doi: 10.1097/AOG.0000000000005496. Epub 2024 Jan 4. PMID 38176019